CLINICAL TRIAL: NCT05853484
Title: FIT4Cirrhotics@Home: Effects of a Home-based Bimodal Lifestyle Intervention in Patients With Liver Cirrhosis Awaiting Orthotopic Liver Transplantation
Brief Title: Home-based Bimodal Lifestyle Intervention in Patients With Liver Cirrhosis Awaiting Orthotopic Liver Transplantation
Acronym: FIT4Cirrhotics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL83612.042.23
Record Dates: First submitted 2023-02-10; First posted 2023-05-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Liver Cirrhosis; Liver Transplant; Complications; Physical Inactivity
MeSH Terms: conditions — Liver Cirrhosis; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home based prehabilitation (Experimental): Participants will be subjected to two training periods of six weeks (or until transplantation) of a semi-supervised home-based bimodal lifestyle program. The bimodal lifestyle program consists of an exercise program combined with nutritional support. The exercise program comprises high intensity interval training and endurance training, combined with peripheral resistance training and breathing exercises
  Interventions: Other: Bimodal lifestyle program

INTERVENTIONS:
Other: Bimodal lifestyle program — Participants will be subjected to two training periods of six weeks (or until transplantation) of a semi-supervised home-based bimodal lifestyle program. The bimodal lifestyle program consists of an exercise program combined with nutritional support. The exercise program comprises high intensity interval training and endurance training, combined with peripheral resistance training and breathing exercises

SUMMARY:
Chronic liver disease eventually results in liver cirrhosis and is associated with an increasing deterioration in patients' physical fitness. As there is currently limited evidence regarding the effects of a home-based exercise program in patients with liver cirrhosis awaiting OLT, and physical frailty rates are particularly high in this patient population, this group has the investigators specific interest. The primary aim of this study is to assess the effect of a semi-supervised home-based bimodal lifestyle program, consisting of interval and endurance training and peripheral resistance training on aerobic capacity in patients with liver cirrhosis awaiting OLT

DETAILED DESCRIPTION:
Rationale: Patients with liver cirrhosis who are on the waiting list for orthotopic liver transplantation (OLT) encounter all key components of physical frailty, i.e., decreased functional capacity, impaired aerobic capacity and sarcopenia, which all lead to fatigue, diminished quality of life, increased hospitalization and pre- and post-transplantation morbidity and mortality. An exercise program in combination with nutritional support has proven to improve all key components of physical frailty and quality of life in various surgical patient populations. Although small studies have demonstrated similar positive effects of exercise training in patients on the waiting list for OLT, to date no large studies supported the effects of exercise training and nutritional support on (the longevity of) the increase in aerobic capacity in OLT patients.

Objective: The primary objective of this study is to assess the effect of a semi-supervised home based bimodal lifestyle intervention on aerobic capacity (measured by VO2 at the Ventilatory anaerobic threshold (VAT) and VO2peak in ml/kg/min) in patients with liver cirrhosis on the waiting list for OLT. Secondary objectives are to evaluate individual patients' responses to the bimodal lifestyle intervention on sarcopenia, anthropometry, functional mobility, quality of life, perceived fatigue, incidence of hepatic encephalopathy, number of unplanned hospital admissions, change in liver frailty index score and change in microbiome composition at six, 12 and 18 weeks, or until transplantation. Finally, the feasibility (participation rate, reasons for non-participation, adherence/compliance, dropout rate, reasons for dropout and adverse event) will be assessed.

Study design: This study is an investigator-initiated, single center, single arm, prospective clinical trial. It will take place at the University Medical Center Groningen, the Netherlands. Eligible patients will participate in the bimodal lifestyle program, which comprises two home-based training periods of six-weeks each (12 weeks training in total, or until transplantation). After 18 weeks (i.e., six weeks after termination of the program) a final assessment will take place to evaluate the longevity of the expected effects of the lifestyle program on predefined study outcomes.

Study population: Adult patients diagnosed with liver cirrhosis and screened for OLT, with a VO2 at the VAT ≤13ml/kg/min and/or VO2peak ≤18ml/kg/min will be screened for potential eligibility. Patients with no contraindications to physical exercise training and the ability to work out on a cycle ergometer can participate in the bimodal lifestyle intervention.

Intervention: Patients will participate in a home-based bimodal lifestyle program. The program comprises semi-supervised high intensity interval and endurance training on an advanced cycle ergometer (Lode Corival Home+ , Lode BV, Groningen, The Netherlands), combined with nutritional support consisting of protein, vitamin and mineral supplementation. Moreover, to improve functional mobility and muscle function patients will perform peripheral resistance training of the large muscle groups of the upper and lower extremities. Finally, to improve respiratory performance after surgery and potentially reduce pulmonary complications, patients will perform breathing exercises. The program will be patient personalized and compromises three training sessions per week. The cycle ergometer used for this program will upload training results of the interval and endurance training sessions to an online platform, enabling remote monitoring of patients' adherence and training progress. Furthermore, a community physical therapist will visit the patient at least weekly to monitor progress and to optimize the training intensity.

Main study parameters/endpoints: The main study parameter/endpoint is the progression in aerobic capacity after 6 weeks. Hereto, before and after the first training period a CPET will performed to determine the difference in VO2 at the VAT and VO2peak in ml/kg/min. A secondary parameter/endpoint of this study is the progression in aerobic capacity after the second training period, and six weeks after termination of the program. Hereto, after 12 and 18 weeks another CPET will be performed. Other secondary parameters/endpoints are the evaluation of differences in sarcopenia, anthropometry, functional mobility, quality of life, perceived fatigue, incidence of hepatic encephalopathy, number of unplanned hospital admissions, change in liver frailty index score and change in microbiome composition at six, 12 and 18 weeks, or until transplantation. Furthermore, postoperative outcomes up to twelve months post-OLT will be collected.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Because the exercise program is situated at home (both the cycle ergometer as the community physiotherapist will come to the patient) the investigators make things as accessible as possible for the patient to participate. Supervision by the physiotherapist during the training sessions is arranged three times in the first week and at least once a week thereafter. At the start of the program a CPET with continuous ECG monitoring will be executed under guidance of trained employees to assess baseline cardiorespiratory fitness, as well as to rule out strain related cardiac ischemia and other contraindications for physical exercise training during the consecutive exercise program. Hence, patient's safety in the exercise program is guaranteed. To minimize the burden of this study, the majority of the visits, withdrawal of blood samples, physical examinations and other study procedures, are combined with regular outpatient clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years;
* Diagnosed with end-stage liver disease / liver cirrhosis (regardless of etiology);
* On the waiting list for OLT;
* VO2 at the VAT ≤13 ml/kg/min and/or VO2peak ≤18 ml/kg/min;
* Speaks the Dutch language;
* Understands the purpose of the study and has given written informed consent to participate in the study.

Exclusion Criteria:

* Experienced a MACE (e.g., myocardial infarction) in the past six months;
* Experienced a cerebrovascular incident in the past six months;
* Medical history of an uncontrolled heart rhythm disorder;
* Hepatic encephalopathy grade 3 or 4;
* Acute liver failure;
* Acute on chronic liver failure;
* Hospitalization at start of the study;
* Non-treated esophageal varices (i.e., variceal eradication endoscopy and/or adequately dosed NSBB);
* MELD score ≥30;
* Not capable of cycling on a cycle ergometer;
* No available community physical therapist in the living area of the patient.
* Patients refusing or unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity | During baseline measurements patients will perform a cardiopulmonary exercise test to determine their baseline aerobic capacity. After 6 weeks of home-based training the cardiopulmonary exercise test will be repeated to reassess their aerobic capacity.
  The main study parameter/endpoint is the change in aerobic capacity after the first six weeks of the FIT4Cirrhotics@Home program, for which the following outcomes will be assessed: VO2 at the VAT (ml/kg/min). A cardiopulmonary exercise test will be performed by participants to determine their aerobic capacity pre-intervention and after six weeks of training.

SECONDARY OUTCOMES:
Ultrasound measurements of muscle thickness | through study completion, an average of 1 year
  Sarcopenia in patients will be assessed by measuring muscle thickness with point-of-care ultrasound before and after the bimodal lifestyle program.
Anthropometry assessment | through study completion, an average of 1 year
  Body mass and height used to calculate the body mass index
Functional mobility assessment | through study completion, an average of 1 year
  30-sec chair-stand test will be performed to assess functional mobility
Quality of Life assessment | through study completion, an average of 1 year
  Questionnaire
Perceived fatigue assessment | through study completion, an average of 1 year
  Questionnaire
Incidence of hepatic encephalopathy assessment | through study completion, an average of 1 year
  Determined using the animal naming test
Number and reasons for intercurrent hospitalizations assessment | through study completion, an average of 1 year
  Number and reasons for intercurrent hospitalizations, with more hospitalizations representing poorer patient outcomes. Minimum hospitalization 0, maximum not predefined.
Liver frailty index score assessment | During through study completion, an average of 1 year and immediately post-intervention
  Determined using https://liverfrailtyindex.ucsf.edu. Scale ranges from 0 - 7 points. A higher score represents a higher risk of clinical frailty.
Microbiome composition assessment | through study completion, an average of 1 year
  By analyzing feces collections
Postoperative outcomes up to 12 months post-OLT assessment | through study completion, and up to 12 months post-OLT assessment
  All surgical relevant postoperative outcomes up to 12 months post-OLT are recorded. Of which, ICU admittance, length of hospital stay, unplanned readmissions, and one-year patient- and graft survival. All displayed as absolute and relative frequencies.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijma AG, Bongers BC, Annema C, Dekker R, Blokzijl H, van der Palen JA, De Meijer VE, Cuperus FJ, Klaase JM. 'Effects of a home-based bimodal lifestyle intervention in frail patients with end-stage liver disease awaiting orthotopic liver transplantation': study protocol of a non-randomised clinical trial. BMJ Open. 2024 Jan 29;14(1):e080430. doi: 10.1136/bmjopen-2023-080430. PMID 38286689